CLINICAL TRIAL: NCT06246968
Title: Does Cryoablation Boost Immune Response Improving the Benefits of Pembrolizumab in Patients With Metastatic or Locally Advanced Triple Negative Breast Cancer?
Brief Title: A Study of Pembrolizumab and Cryoablation in People With Breast Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-390
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Breast Cancer; Breast Cancer; Breast Cancer Stage IV; Triple Negative Breast Cancer; Triple Negative Breast Neoplasms; Metastatic Triple-Negative Breast Carcinoma; Locally Advanced Breast Cancer; Locally Advanced Triple-Negative Breast Carcinoma
Keywords: metastatic TNBC; metastatic triple negative breast carcinoma; metastatic breast cancer; breast cancer; breast cancer stage IV; triple negative breast cancer; pembrolizumab; cryoablation; Memorial Sloan Kettering Cancer Center; 23-390; locally advanced breast cancer; locally advanced triple negative breast carcinoma; locally advanced triple negative breast cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — pembrolizumab; Cryosurgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Pembrolizumab + Cryoablation (Experimental): Participants will have a diagnosis of metastatic triple negative breast cancer or locally advanced inoperable triple negative breast cancer. Participants will be randomized 2 (cryoablation arm): 1 (no cryoablation arm).
  Interventions: Drug: Pembrolizumab; Device: Cryoablation
- Pembrolizumab (Active Comparator): Participants will have a diagnosis of metastatic triple negative breast cancer or locally advanced inoperable triple negative breast cancer. Participants will be randomized 2 (cryoablation arm): 1 (no cryoablation arm).
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Participants will receive Pembrolizumab as part of standard of care treatment.
Device: Cryoablation — Cryoablation is a type of thermal ablation that is a minimally invasive alternative technique to surgical resection.
  Arms: Pembrolizumab + Cryoablation

SUMMARY:
Participants will have a confirmed diagnosis of metastatic breast cancer and will receive pembrolizumab in combination with cryoablation OR pembrolizumab alone. Participants will be randomly assigned.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age
* Confirmed histologic diagnosis of metastatic TNBC
* 1 site amenable cryoablation of at least 1.5 cm in size as determined by an Interventional Radiologist. Eligible cryoablation sites include (but not limited to) soft tissue, liver, lung, and bone as determined by an Interventional Radiologist to be safest and most feasible.
* Physically fit (clinically eligible) to undergo cryoablation as per usual clinical practice
* Per clinical guidelines, women of childbearing age should use effective contraception during treatment with pembrolizumab and for at least 4 months after the last dose of the drug, which will be assessed and monitored by, and the responsibility of, the patient's medical oncologist (not study investigators or research team) as pembrolizumab is standard of care. Memorial Sloan Kettering Cancer Center Pregnancy Standards will be followed prior to cryoablation. That is, female patients that are 11-50 years of age and of childbearing potential will undergo a pregnancy test within 2 weeks (15 days) before cryoablation. Pregnancy test will not be required in patients with bilateral oophorectomy, bilateral salpingectomy, bilateral salpingectomy-oophorectomy, hysterectomy, menopause (no menses ≥ 1 year prior to treatment or after completion of all treatment), or surgical sterilization (i.e. tubal ligation or blockage), with documentation of permanent exemptions in CIS ("Pregnancy Testing Exemption").
* Pembrolizumab therapy (200 mg every 3 weeks) planned as part of standard of care as first, second, or third line of therapy

  * Eligible for PD-1 inhibitor per the patient's medical oncologist, with planned treatment with PD-1 inhibitor per the patient's medical oncologist. Additional systemic therapy is per the patient's medical oncologist. The following systemic therapy will be accepted (the timing of the systemic therapy relative to pembrolizumab and cryoablation is not restricted):

    * Capecitabine (Xeloda, available as a generic drug)
    * Carboplatin (Paraplatin, available as a generic drug)
    * Cisplatin (Platinol, available as a generic drug)
    * Cyclophosphamide (Cytoxan, available as a generic drug)
    * Docetaxel (Taxotere)
    * Doxorubicin (Adriamycin, available as a generic drug)
    * Pegylated liposomal doxorubicin (Doxil)
    * Epirubicin (Ellence, available as a generic drug)
    * Eribulin (Halaven)
    * Fluorouracil (5-FU, Adrucil, available as a generic drug)
    * Gemcitabine (Gemzar, available as a generic drug)
    * Ixabepilone (Ixempra)
    * Methotrexate (available as a general drug)
    * Nab-paclitaxel (Abraxane)
    * Paclitaxel (Taxol, available as a generic drug)
    * Vinorelbine (Navelbine, available as a generic drug)

Exclusion Criteria:

* Patient not eligible for PD-1 inhibitor per the patient's medical oncologist
* No disease amenable for cryoablation
* Pembrolizumab therapy not planned as part of standard of care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2027-01-29 (Estimated); Study Completion 2027-01-29 (Estimated)

PRIMARY OUTCOMES:
Change in CD4-PD1 from baseline to post-cryoablation | 6 weeks after cryoablation
  Assess changes in CD4-PD1 in the blood after cryoablation in patients with metastatic or locally advanced triple negative breast cancer (TNBC).

CONTACTS AND LOCATIONS:
Overall Officials: Yolanda Bryce, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Cancer Center at Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (Limited Protocol Activities ), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All protocol activites), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activites), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org